CLINICAL TRIAL: NCT02335320
Title: Qualification of Point-of-Care Assays for Management of HCV Patients
Acronym: ANRS HC POC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS HC POC
Record Dates: First submitted 2014-11-24; First posted 2015-01-09 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Hepatitis C
Keywords: VHC; IL28-B; point of care
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute or chronic HCV infection can lead to liver complications, including liver failure, cirrhosis or liver cancer. For patients with hepatitis C infection, the major clinical question remains the terms of treatment initiation. In Europe, new treatments are available since the approval of three direct acting antivirals. However with the high cost of these treatments, they are currently only available for critically ill patients. Other molecules are currently in advanced clinical development phases. The use of clinical predictors remains relevant for the selection of a suitable treatment for each patient, in particular to limit the adverse effects and reduce costs. Currently the quantification of viral load is a measure of response to treatment; with the recommendation to stop treatment in patients who fail to achieve an undetectable level of viral load. Genetic factors have also been identified as predictors of response to treatment, in particular polymorphisms of the IL-28B gene. Genotyping of this gene is currently performed using classical PCR amplification applied to DNA extracted from blood, with a time to result of 2-3 weeks. We propose in this protocol to test a non-invasive method and rapid test for IL-28B genotype which could be used for point of caring testing, and ultimately better patient management.

This is a monocenter, cross-sectional study among HCV chronic patients. The study will be conducted in 250 HCV patients, all viral genotypes combined, at Cochin Hospital (Paris, France).

Objectives The principal objective is to assess the accuracy of the newly developed Point-of-Care genotyping assay (Genedrive® IL-28B Assay) to detect in HCV patients the genotype CC versus non CC (i.e. CT and TT) against the TaqMan Allelic Discrimination Assay as gold standard.

The secondary objective is to assess the concordance between the genotype results of the Genedrive and the gold standard regarding the three genotypes CC, CT and TT.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Patients diagnosed with hepatitis C (all viral genotypes).
* Patient already treated or recommended to start antiviral therapy against hepatitis C virus or currently undergoing antiviral therapy.
* Patients who consented to IL-28B genotyping in the course of their usual follow-up by conventional PCR standard method.
* Patients affiliated to social security.
* Informed consent must be obtained for all subjects prior to study entry.

Exclusion Criteria:

* A person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV chronic patients (all viral genotypes)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
proportion of patients with genotype IL-28B C/C versus IL-28B non C/C patients | D1
  The study is based on the comparison of the genotyping results for SNP rs1297860 (IL-28B gene) between the Genedrive® assay and the gold standard assay.

SECONDARY OUTCOMES:
proportion of patients of whom the genotype results are identical between the index test and the gold standard test. | D1
  For secondary endpoints the three genotypes (C/C, C/T, T/T) are considered

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Cochin Saint-Vincent de Paul, Paris, France